CLINICAL TRIAL: NCT06995885
Title: Development of an Interview-Informed Timeline Follow-Back (TLFB) for Opioid Use in the Era of Fentanyl
Status: Enrolling by invitation | Type: Observational
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10002297; 002297-DA
Record Dates: First submitted 2025-05-28; First posted 2025-05-30 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12-02

CONDITIONS: Substance Use Disorders (SUDs)
Keywords: People who use opioids (PWUOs); Opioids; Timeline Follow-Back (TLFB)
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- People who use opioids (PWUOs): Past 30-day use of an opioid obtained in a nonmedical context (i.e., not from a pharmacy or in a healthcare setting)

SUMMARY:
Background:

A Timeline Follow-Back (TLFB) is a tool that helps researchers track how much of a substance a person uses. Different versions of the tool are used to track the use of alcohol, cigarettes, and cannabis. But there is no TLFB to track a person s use of nonmedical opioids. (These are opioids not obtained from a medical source; they may also be called "street" opioids.) Researchers are creating an Opioid TLFB (OpiTLFB) that asks better questions and records more useful answers to identify what kinds of nonmedical opioids people are using.

Objective:

To test a new research tool to track a person's use of nonmedical opioids.

Eligibility:

People aged 18 years or older who used a nonmedical opioid within the past 30 days.

Design:

Participants will have 1 study visit at a clinic in Baltimore, Maryland. The visit will take 1 to 4 hours.

Participants will sit at a computer with a researcher and fill out a calendar. They will record their use of opioids each day for the past 30 days. They will be asked what the drugs were called and what they looked like. This task might take 30 minutes.

Participants will be interviewed. The researcher will ask about their experiences getting opioids from friends, dealers, or other sources; how the experience of getting opioids has changed over time; and about any changes they have noticed across different areas of Baltimore. Researchers will ask how the OpiTLFB could be easier to fill out and how it could provide more useful information. This task might take 30 minutes.

Participants will provide a urine sample.

DETAILED DESCRIPTION:
Study Description:

Observational, on-site study for the purpose of instrument development. Currently used assessments of recent opioid use do not reflect the current market for street opioids. This protocol will use semistructured interviews (supplemented with results from comprehensive toxicology of approximately 1,200 analytes in urine) to develop a workable typology of the current street-opioid market in the Baltimore region, and a TLFB calendar that asks germane questions and offers usable response options for products and amounts.

Objectives:

1. To conduct semistructured interviews with people who use opioids (PWUOs) in the Baltimore area about their recent opioid use, for development of a TLFB instrument that assesses use in terms that accord with the current conditions of the market.
2. To perform comprehensive toxicology testing so that an appearancedriven and effect-driven typology of street opioids can be tentatively mapped onto their likely contents.

Endpoints:

1. At least three consecutive respondents (after an initial minimum of 25 respondents) for whom the OpiTLFB needs no further modification to capture their pattern of opioid use.
2. Associations between OpiTLFB indices (name, physical appearance, and effects of product) and urine-toxicology results.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to participate in this study, an individual must meet the following criteria:

1. Age 18 years or older
2. Past 30-day use of an opioid obtained in a nonmedical context (i.e., not from a pharmacy or in a healthcare setting)
3. Able to understand and communicate in written and spoken English.

   Justification: Initial development of the OpiTLFB requires strong, unmediated communication between the study team and the participants. Further development and modification for non-English-speaking interviewees is best undertaken as a separate project when the OpiTLFB is ready for use.
4. Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

1. Any medical, psychiatric, or social conditions that the investigators believe would make participation in this protocol not in the best interest of the participant.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We may enroll participants in this protocol from the pool that screens for other protocols at the NIDA IRP. We may also advertise for this protocol directly. If we decide to launch an ad campaign for this specific protocol, we will primarily recruit in the Baltimore metro area. We may also recontact previous participants from NIDA IRP studies who have expressed interest in participating in future NIDA studies and agreed to such recontact. Additionally, study team members attend events hosted by the Office of the Clinical Director to engage with local community partners. This includes clinics, treatment facilities, medical facilities, advocacy groups, and local businesses. We conduct outreach at community events/locations such as health expos, festivals, and other local venues. During these events, we display and offer approved recruitment materials.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
At least three consecutive respondents (after an initial minimum of 25 respondents) for whom the OpiTLFB needs no further modification to capture their pattern of opioid use. | 6-24 months
  Existing TLFB measures assess opioid use in terms that no longer match what PWUOs can actually obtain. This hampers both baseline characterization and quantification of opioid-use changes in study participants.
Associations between OpiTLFB indices (name, physical appearance, and effects of product) and urine-toxicology results. | 6-24 months
  This will help ensure that our typology of street opioids reflects real and consistent differences in product composition.

CONTACTS AND LOCATIONS:
Overall Officials: David H Epstein, Ph.D., Principal Investigator — National Institute on Drug Abuse (NIDA)
Locations (1):
- National Institute on Drug Abuse, Baltimore, Maryland, United States